CLINICAL TRIAL: NCT07187102
Title: Ultrasonographic Response to Cervical and Upper Thoracic SNAG in Treatment of Chronic Medial Epicondylitis, Randomized Clinical Trial
Brief Title: Ultrasonographic Response to Cervical and Upper Thoracic SNAG in Medial Epicondylitis, Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sahar Mowad Abdelmutilibe, faculty of physical therapy , beni suef university, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/07092025/Ahmed
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Medial Epicondylitis
Keywords: mobilization , SNAG , medial epicondylitis
MeSH Terms: conditions — Elbow Tendinopathy

STUDY DESIGN:
Intervention Model Description: one group receive SNAG plus traditional treatment second group receive traditional treatment
Masking Description: Open Label - both participants and investigators will be aware of the intervention received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participants will receive the physiotherapy SNAG plus traditional treatment program (4weeks, supervised sessions 3 times per week )
  Interventions: Other: SNAG ( sustained natural apopheseal glide )
- control group (Other): Participants will receive the physiotherapy traditional treatment program (4weeks, supervised sessions 3 times per week )
  Interventions: Other: SNAG ( sustained natural apopheseal glide )

INTERVENTIONS:
Other: SNAG ( sustained natural apopheseal glide ) — SNAG : type of mobilization of vertebral coulmn

SUMMARY:
Aim of the work :

1. To detect if there is any change would occur in the neovascularity and echogenicity after using cervical and upper thoracic SNAG or not in ME patients.
2. To find the effect of cervical and upper thoracic SNAG on pain, function of upper extremities, grip strength in ME comparing with traditional treatment alone

DETAILED DESCRIPTION:
medial epicondylitis(ME) of the elbow is a condition characterized by aggravation of pain in the outer part of the elbow during active wrist flexion , and presentation of pain on direct palpation of the medial epicondyle, or proximal muscle belly . Biomechanical and sensorimotor deficits can occur and adversely impact upper extremity function .These functional deficits may interfere with occupational tasks and activities of daily living The study's results: Measuring the changes that will be produced by using therapeutic growth of the cervical and thoracic vertebrae on the pathological changes that persist in the tendons of the tens of the tibialis cruciate ligaments in detecting excess weight resulting from the disease of the middle epicondyle, such as increased blood vessels in the tendon and decreased echogenicity of the tendon, in addition to measuring the changes that occurred in the extent of pain sensation and the extent of functional performance of the shoulder and elbow joints. Patients will be directly selected jointly according to the patient's specifications for the research and written consent will be obtained from the patient after a detailed explanation of the research steps and what is required of him. The vocal function of the tendon will be evaluated, with the exception of functional pain of the successful upper extremity and the strength of the hand muscles before and after the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 35 to 50 years old in both sexes.
* Patients with LE that diagnosed by orthopedist.
* Pain onset is more than 3 months appear primarily with use or rest or in both, also , it appear with deep palpation of the medial epicondyle .

Exclusion Criteria:

* • Rheumatoid Arthritis .

  * Skin infection.
  * History of previous elbow surgery.
  * Any pathology in the shoulder joint.
  * Neurologic deficit in upper extremity.
  * Cervical disc prolapse and radiculopathy C5,6.
  * Dislocation of elbow joint.
  * Recent fractures of upper extremity.
  * Arthrosis of the radiohumeral joint.
  * Osteochondritis dissecans.
  * Osteonecrosis.
  * Plica synovialis.
  * Participants receiving other treatment, in the form of physical therapy or medication, for the duration of the study that may interfere with the results of this study.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in hypervascularity and hypoechogencity measured by colour sonography ( grade 1: grade 4) | 2 months
  Change in hypervascularity and hypoechogencity measured by colour sonography ( grade 1: grade 4)
Change in shoulder disability measured by DASH SCALE and elbow disability by PRTEE scale ) | 2 MONTHS
  Change in shoulder disability measured by DASH SCALE and elbow disability by PRTEE scale )
Change in pain intensity measured by Visual Analogue Scale (VAS, 0-10 points) | 2 months
  Change in pain intensity measured by Visual Analogue Scale (VAS, 0-10 points)
Change in grip muscle strength measured by hand held dynamometer points | 2 months
  Change in grip muscle strength measured by hand held dynamometer points

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Beni-Suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No
"No, there is no plan to make individual participant data (IPD) available to other researchers due to privacy concerns and institutional restrictions."